CLINICAL TRIAL: NCT03578354
Title: Prospective, Randomized, Placebo-controlled, Phase 2 Study of 4-aminopyridine, Atenolol, or Placebo in the Treatment of Patients With Vestibular Migraine
Brief Title: 4-Aminopyridine, Atenolol, or Placebo in Patients With Vestibular Migraine
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Funding not acquired
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Responsible Party: Principal Investigator, Richard Lewis, Associate Professor, Otolaryngology and Neurology; Director, Jenks Vestibular Laboratory, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Pending
Record Dates: First submitted 2018-05-31; First posted 2018-07-06 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Vestibular Migraine; Migraine Disorders; Vestibular Diseases
MeSH Terms: conditions — Migraine Disorders; Vestibular Diseases | interventions — 4-Aminopyridine; Atenolol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- 4-AP (Experimental): 15 mg 4-aminopyridine twice daily
  Interventions: Drug: 4-aminopyridine
- Atenolol (Experimental): 25 mg atenolol twice daily
  Interventions: Drug: Atenolol
- Placebo (Placebo Comparator): Masked placebo twice daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: 4-aminopyridine — an oral drug to be swallowed
  Arms: 4-AP
Drug: Atenolol — an oral drug to be swallowed
  Arms: Atenolol
Other: Placebo — a masked placebo to be swallowed
  Arms: Placebo

SUMMARY:
This phase 2 randomized study will be used to test the efficacy of 4-aminopyridine (4AP) or atenolol to reduce severity and frequency of vestibular and headache symptoms of vestibular migriane sufferers. Blinded study drug will be taken by mouth twice a day for 14 weeks on study.

ELIGIBILITY:
Inclusion Criteria:

* Severe vestibular migraine (VM)

Exclusion Criteria:

* Neurologic or otologic disease other than VM
* Psychiatric illness requiring medication
* Medical illness including cancer, coronary artery or cerebrovascular disease
* Known allergy to one of the test medications
* Contraindication to use of one of the test medications - asthma, symptomatic hypotension, history of seizures
* Taking migraine prophylactic medication or vestibular suppressants.
* Pregnant or breast feeding women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-01 (Estimated); Primary Completion 2023-01 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Change in Dizziness Handicap Score | 14 weeks
  Dizziness Handicap Inventory (DHI) will be compared pre- and post- study drug treatment

SECONDARY OUTCOMES:
Change in number of dizziness episodes | 14 weeks
  Incidence of dizziness episodes will be compared pre- and post- study drug treatment
Change in motion sickness susceptibility | 14 weeks
  Motion sickness susceptibility questionnaire (MSSQ) will be compared pre- and post- study drug treatment. MSSQ is reported as a scale (0 - 100) with 0 being no or very little experience of motion sickness, and 100 being very frequent experience of motion sickness.
Change in roll tilt perceptual threshold | 14 weeks
  Rolt tilt perceptual thresholds will be compared pre- and post- study drug treatment
Change in vestibulo-ocular reflex (VOR) time constant | 14 weeks
  Standard low-frequency rotational testing to measure VOR will be compared pre- and post- study drug treatment
Change in number of migraine episodes | 14 weeks
  Incidence of migraine episodes will be compared pre- and post- study drug treatment
Change in Headache Impact Test (HIT) score | 14 weeks
  Headache Impact Test (HIT) will be compared pre- and post- study drug treatment
Change in quality of life score | 14 weeks
  Quality of life will be measured using 36-Item Short Form Health Survey (SF-36) questionnaires and compared pre- and post- study drug treatment. The SF-36 consists of 8 sub-scores. Each score is reported as a scale (0 - 100) with 0 being maximally disabled and 100 having no disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States